CLINICAL TRIAL: NCT04510987
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of a Single Oral Dose of 25 mg BAY 2433334 in Male and Female Participants With Different Stages of Renal Impairment (Including on Dialysis), as Compared to Age, Gender and Weight Matched Participants in a Single-center, Non-randomized, Non-controlled, Non-blinded, Group Stratification Design Study.
Brief Title: Study to Assess the Safety, Tolerability, Effects on the Body, Absorption, Distribution and Elimination of 25 mg BAY2433334 in Renal Impairment Including Renal Replacement Therapy ("Dialysis")
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19771; 2020-000626-25 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-08-12 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Prevention of Thromboembolic Events
Keywords: Renal impairment; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Treatment 1 (Experimental): Participants in Groups 1-4 and Group 6 will receive a single dose of BAY2433334 on one occasion. Participants in Group 5 will receive a single dose of BAY2433334 on a dialysis-free day.
  Interventions: Drug: BAY2433334 single dose in treatment groups 1-4 and 6 as well as on the dialysis free day of treatment 5
- Experimental: Treatment 2 (Experimental): Participants in Group 5 will receive a single dose of BAY2433334 on a day with dialysis treatment.
  Interventions: Other: BAY2433334 on dialysis treatment day

INTERVENTIONS:
Drug: BAY2433334 single dose in treatment groups 1-4 and 6 as well as on the dialysis free day of treatment 5 — Tablet, oral
  Arms: Experimental: Treatment 1
Other: BAY2433334 on dialysis treatment day — Tablet, oral
  Arms: Experimental: Treatment 2

SUMMARY:
BAY2433334 is under clinical development for prevention of complications in diseases such as heart attack, irregular heart beat or stroke which can arise by formation of blood clots elsewhere in the body and travels through the blood stream to plug another vessel. Renal impairment which co-occurs in elderly and patients with heart attack, irregular heart beat or stroke is a common condition in which the kidneys are not filtering the blood as well as they should. The goal of the study is to learn more about the safety of BAY2433334, how it is tolerated and the way the body absorbs, distributes and gets rid of the study dug given as a single oral dose of 25 mg tablet in participants with renal impairment and healthy participants matched for age-, gender-, and weight.

ELIGIBILITY:
Inclusion Criteria:

* All participants: ≥18 years, male or female (non-WOCBP only), BMI 18-35 kg/m² (inclusive); no increased risk of bleeding or common causes of bleeding, no liver dysfunction; no CYP3A4 inhibitors/inducers;
* Participants with reduced kidney function including those on kidney replacement therapy ("dialysis"): stable disease stratified by renal function (mild, moderate, severe, ESRD), no recent cardiovascular events;
* Age-, gender- and weight-matched participants: normal kidney function, stable and well controlled hypertension and dyslipidemia acceptable, no medications influencing the coagulation system.

Exclusion Criteria:

Subjects with renal impairment

* Acute renal failure or active nephritis.
* Known impaired hepatic function.
* History of definite myocardial infarction or cerebrovascular accident within the six months prior to the screening visit.
* History of vascular surgery or intervention (e.g., coronary artery bypass, percutaneous transluminal angioplasty etc.) less than 6 months prior to dosing.
* Congestive heart failure of New York Heart Association grade III or IV, severe arrhythmia requiring antiarrhythmic treatment.
* Any other disease or condition which could influence the physiological metabolic turnover (e.g., endocrine diseases, severe infections).

Age-, gender, weight matched subjects

- History of relevant diseases of vital organs or systems (e.g., of the central nervous system or other systems or organs) with the exception of mild, well controlled hypertension, dyslipoproteinemia and thyroid disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose until 96 hours after dosing
  maximum observed drug concentration in measured matrix after single dose administration
AUC | Pre-dose until 96 hours after dosing
  area under the concentration vs. time curve from zero to infinity after single (first) dose AUC(0-tlast) and AUC(0-tlast)u will be used as primary variables if mean AUC(tlast-∞) >20% of AUC
Cmax,u | Pre-dose until 96 hours after dosing
  maximum unbound drug concentration in plasma after single dose administration
AUCu | Pre-dose until 96 hours after dosing
  area under the unbound plasma concentration vs time curve from zero to infinity after single (first) dose AUC(0-tlast) and AUC(0-tlast)u will be used as primary variables if mean AUC(tlast-∞) >20% of AUC

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | Up to 3 days after last study medication

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.